CLINICAL TRIAL: NCT06002035
Title: The Role and Mechanism of Vitamin D in Recurrent Spontaneous Abortion Based on Maternal Fetal Interface Immune Tolerance
Brief Title: Study on Clinical Value of Vitamin D in Recurrent Spontaneous Abortion
Status: Completed | Type: Observational
Sponsor: Jianmei Xia (Other)
Responsible Party: Sponsor-Investigator, Jianmei Xia, Deputy Chief Physician, First People's Hospital of Hangzhou
Organization: First People's Hospital of Hangzhou (Other)
Other Study IDs: 2023002
Record Dates: First submitted 2023-07-31; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Vitamin D Deficiency; Recurrent Spontaneous Abortion
MeSH Terms: conditions — Vitamin D Deficiency; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- patients without spontaneous abortion(SA0): The patients with VD deficiency or insufficiency take 30 drops (relative to 1ml) once a day, directly into the mouth or with complementary foods added.
  Interventions: Dietary Supplement: Binom Vitamin D drops
- patients with a spontaneous abortion(SA1): The patients with VD deficiency or insufficiency take 30 drops (relative to 1ml) once a day, directly into the mouth or with complementary foods added.
  Interventions: Dietary Supplement: Binom Vitamin D drops
- patients with RSA (SA2 and above): The patients with VD deficiency or insufficiency take 30 drops (relative to 1ml) once a day, directly into the mouth or with complementary foods added.
  Interventions: Dietary Supplement: Binom Vitamin D drops

INTERVENTIONS:
Dietary Supplement: Binom Vitamin D drops — Take 30 drops (relative to 1ml) once a day, directly into the mouth or with complementary foods added

SUMMARY:
The observational study is to compare vitamin D deficiency and related indicators among different spontaneous abortions in describe female reproductive health.The main question aim to answer is: the possible pathogenesis of recurrent spontaneous abortion caused by vitamin D.

Participants, who visit the RSA specialty clinic, will provide medical history information, regularly exam based on the condition, following up on pregnancy status.Participants will be asked to supply vitamin D preparation and do moderate exercise outdoors, comparing the effect after treatment.

DETAILED DESCRIPTION:
Examinations include uterine artery resistance parameter S/D, some embryonic chromosomes tested voluntarily, plasma VD content and the level of anticardiolipin antibody.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of patients without spontaneous abortion;
* Clinical diagnosis of patients with a spontaneous abortion;
* Clinical diagnosis of patients with recurrent pontaneous abortions;

Exclusion Criteria:

* Patients with chromosomal abnormalities in RSA couples, such as balanced translocation;
* Patients who take VD preparations or related VD supplements within 3 months before treatment;
* Patients with a combination of certain malignant tumors and severe mental illness.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women of childbearing age visited the RSA specialty clinic of Hangzhou First People's Hospital from January 2021 to June 2023, conducting a prospective clinical study.
Sampling Method: Probability Sample
Enrollment: 1421 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Rate of the effect of vitamin D supplementation on adverse pregnancy outcomes1 | average of 1 year
  Through outpatient follow-up, follow-up and inpatient information, pregnancy outcomes are classified according to Williams obstetrics, such as empty sac which refers to the absence of a fetal sac or embryo bud (the amniotic sac is empty).
Rate of the effect of vitamin D supplementation on adverse pregnancy outcomes2 | average of half of a year
  Through outpatient follow-up, follow-up and inpatient information, pregnancy outcomes are classified according to Williams obstetrics, such as biochemical pregnancy which refers to the phenomenon where the sperm and egg combine but fail to return to the uterus for implantation, leading to miscarriage along with menstruation.
Rate of the effect of vitamin D supplementation on adverse pregnancy outcomes3 | average of half of a year
  Through outpatient follow-up, follow-up and inpatient information, pregnancy outcomes are classified according to Williams obstetrics, such as loss of fetal heart rate which refers to the cessation of fetal heartbeat during pregnancy leading to miscarriage.
Rate of the effect of vitamin D supplementation on adverse pregnancy outcomes4 | average of half of a year
  Through outpatient follow-up, follow-up and inpatient information, pregnancy outcomes are classified according to Williams obstetrics, such as spontaneous miscarriage in large months (greater than 12 weeks but less than 28 weeks) which refers to the cause of fetal death in the uterus, vaginal bleeding or flowing and abdominal pain leading to miscarriage.
Rate of the effect of vitamin D supplementation on adverse pregnancy outcomes5 | average of half of a year
  Through outpatient follow-up, follow-up and inpatient information, pregnancy outcomes are classified according to Williams obstetrics, such as failure of fetal heart rate which the inability of the fetus to detect heartbeat leading to miscarriage.

SECONDARY OUTCOMES:
The difference of age in different number of spontaneous abortions | one day
  Record patients' age through initial visit.
The difference of BMI in different number of spontaneous abortion | one day
  Record patients' height and weight through initial visit, and then calculate according to BMI formula.
The difference of uterine artery resistance parameter S/D in different number of spontaneous abortions | dynamic monitoring, average of half of a year
  Use a three-dimensional ultrasound diagnostic instrument(GEVoluson-E10 or E8, USA) with a frequency of 5-9 MHz intracavity probe (non pregnancy) or 3-7 MHz abdominal probe (pregnancy) to examine bilateral S/D. Unpregnant patients were in mid luteal phase(5-7 days after ovulation), while pregnant patients were at 10 weeks of pregnancy.
The abnormality of some embryonic chromosomes tested voluntarily in spontaneous abortions | a month
  use SNP gene chips to detect the embryonic chromosomes in spontaneous abortion; extract the genomic DNA of aborted embryo tissue, perform whole genome chromosome detection and determine whether the corresponding fragment or site is abnormal.
The change of plasma VD content in spontaneous abortions before and after supplying vitamin D | average of 1 year
  VD content was detected by liquid chromatography-tandem mass spectrometry using DISIGNS reagent. Dynamically monitor plasma VD at least twice every two months before and after treatment, and monitor early, mid, and late pregnancy each once after conception.
The change of the level of plasma anticardiolipin antibody in spontaneous abortions before and after supplying vitamin D | average of 1 year
  ACA level was detected by enzyme-linked immunosorbent assay using EUROIMMUN reagent. dynamically monitor plasma anticardiolipin antibody at least twice every two months before and after treatment, and monitor early, mid, and late pregnancy each once after conception.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmei Xia, Study Director — First People's Hospital of Hangzhou
Locations (1):
- Jianmei Xia, Hangzhou, Zhejiang, China